CLINICAL TRIAL: NCT01132638
Title: Evaluation of Complete Remission of Erosive Gastroesophageal Reflux Disease Following Four-week Treatment With Pantoprazole Magnesium 40 mg Versus Esomeprazole 40 mg With Eight-week Extension Treatment in Non-responding Patients - Multicenter, National, Prospective, Randomized, Double-blind, Parallel-group, Phase III
Brief Title: Pantoprazole Magnesium 40 mg Versus Esomeprazole 40 mg in Patients With Erosive Gastroesophageal Reflux Disease
Acronym: PAMES 0109
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PZ-9999-401-BR; U1111-1130-9255 (Registry Identifier: WHO)
Record Dates: First submitted 2010-05-21; First posted 2010-05-28 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: GERD
Keywords: Gastroesophageal; Pantoprazole; erosive; Erosive GERD grades A-D, acc. to Los Angeles classification
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Magnesium Pantoprazole (Active Comparator)
  Interventions: Drug: Magnesium Pantoprazole
- Magnesium Esomeprazole (Active Comparator)
  Interventions: Drug: Magnesium Esomeprazole

INTERVENTIONS:
Drug: Magnesium Pantoprazole — 1 capsule daily, 40 mg, orally, 30 minutes before breakfast
  Arms: Magnesium Pantoprazole
Drug: Magnesium Esomeprazole — 1 capsule daily, 40 mg, orally, 30 minutes before breakfast
  Arms: Magnesium Esomeprazole

SUMMARY:
The aim of this trial is to evaluate the complete remission of erosive gastroesophageal reflux disease with pantoprazole magnesium 40 mg once daily versus esomeprazole 40 mg once daily during four-week treatment with an extension treatment for non-responding patients. The study includes a baseline period up to 14 days and a treatment period of either 4 weeks (28 -2 + 5 days), or 8 weeks depending on the cure of esophagitis due to gastroesophageal reflux. The study will provide further data on safety and tolerability of pantoprazole magnesium.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study with signature on Informed Consent Form (ICF) prior to specific protocol procedures
* Patients of any race
* On outpatient treatment
* History of frequent symptom crises related to GERD within the last 3 months (at least a frequency of twice a week, for about four to eight weeks)
* Diagnosis of erosive esophagitis (grade A to D, according to Los Angeles Classification)
* In good health condition, except GERD symptoms
* Able to follow the protocol directions and to complete daily the questionnaire ReQuest™ throughout the study

Exclusion Criteria:

* Gastrointestinal disorder, even when related to chlorhydropeptic disorders: Barret's esophagus, peptic ulcer, Zollinger-Ellison syndrome and pyloric stenosis
* Previous history of surgery to reduce acid secretion, or other upper gastrointestinal tract surgeries (excepting polypectomy and cholecystectomy)
* At initial endoscopy presenting complicated disorders due to erosive esophagitis: obstructive esophageal stenoses, Schatzki ring, esophageal diverticulum, esophageal varices, achalasia and hiatal hernia
* Pregnant women or during nursing period
* Proton Pump Inhibitors (PPIs) within the last 10 days prior to start of the study
* Triple therapy based on PPIs to eradicate H. pylori within the last 28 days prior to start of the study
* H2-blockers, sucralfate and prokinetics within the last 7 days prior to start of the study
* Systemic glucocorticoids and/or nonsteroidal anti-inflammatory drugs (including COX-2 inhibitors) for more than 3 consecutive days a week, within the last 28 days prior to start of study, with exception of regular intake of acetyl salicylic acid in dosages of up to 163 mg/day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Comparatively evaluation of the clinical efficacy of pantoprazole magnesium and esomeprazole in the treatment of patients with erosive gastroesophageal reflux disease (GERD), considering the proportion of patients in complete remission. | After 4 treatment weeks
  A patient is considered at complete remission if he/she achieved symptoms relief and confirmed endoscopic healing at treatment end. A patient achieves symptoms relief if Reflux Questionnaire-GI score ((ReQuest™) stays below 1,73 for at least the three last consecutive treatment days, that can occur at visit V2 or visit V3 for those that did not achieve complete remission at V2 and repeated the treatment for 4 weeks more.

SECONDARY OUTCOMES:
Treatments comparative evaluation for DRGE ReQuest™-GI and -WSO scores change with respect to baseline measured | After 4 and 8 treatment weeks
Treatments comparative evaluation for the time interval from treatment start to the beginning of symptoms relief
Treatments comparative evaluation for endoscopic healing rate | After 4 and 8 treatment weeks

CONTACTS AND LOCATIONS:
Locations (9):
- Brazil (9):
  - Investigational site, Belo Horizonte/MG
  - Investigational site, Curitiba/PR
  - Investigational site, Goiânia/GO
  - Investigational site, Porto Alegre/RS
  - Investigational site, Ribeirão Preto/SP
  - Investigational site, Rio de Janeiro/RJ
  - Investigational site, Salvador/BA
  - Investigational site, Santo André/SP
  - Investigational site, São Paulo/SP

REFERENCES:
- [Derived] Moraes-Filho JP, Pedroso M, Quigley EM; PAMES Study Group. Randomised clinical trial: daily pantoprazole magnesium 40 mg vs. esomeprazole 40 mg for gastro-oesophageal reflux disease, assessed by endoscopy and symptoms. Aliment Pharmacol Ther. 2014 Jan;39(1):47-56. doi: 10.1111/apt.12540. Epub 2013 Oct 29. PMID 24299323